CLINICAL TRIAL: NCT05446415
Title: Evaluation of L-Cell Activity in the Small Intestine as Biliopancreatic Loop Extension in Obese Patients With DM2 Submitted to Roux-en-Y Gastric Bypass
Brief Title: L-Cell Activity in Small Intestine as Biliopancreatic Loop in Obese Patients With DM2 Submitted to RYGBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marco Aurélio Santo, Principal investigator, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 65854317800000068
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Severe Obesity; Type 2 Diabetes Mellitus in Obese
Keywords: Roux-en-Y gastroplasty; Immunohistochemistry; L cell; GLP-1; PYY; type 2 diabetes
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2 | interventions — Glucagon-Like Peptide 1; Peptide YY; peptide YY (3-36)

STUDY DESIGN:
Intervention Model Description: Roux-en-Y bypass gastroplasty (GDYR) by laparoscopy, with production of a gastric pouch with a volume between 30 and 50 ml, with a biliopancreatic loop measuring 100 (G1) and 200 cm (G2), anastomosis of the alimentary loop of 100 cm in the groups G1 and G2.
  Immunohistochemistry analysis assays were made from intestinal biopsies in 3 segments: gastrointestinal anastomosis (GEA = Point A), enteroenteral anastomosis (EEA = Point B ) and (Ileocecal valve =Point C).
  Expression and secretion of GLP-1 and PYY3-36, incretins hormones by Lcells.
Masking Description: Study is randomized by the RedCap program, until the time of surgical intervention Researcher and Participant do not know the model. On the day of the Bariatric Surgery, the Participant's data are placed in the program to generate randomization, after the result, only the Researcher and team will know the model chosen by the program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective analisys (Other): Immunohistochemical assays : biopsy sampled from each site was immediately fixated and then embedded in paraffin, cut in thin slide sections and dewaxed. Subsequently, antigen retrieval was performed, with incubations with (1) specific primary antibodies, (2) a second layer of antibodies and (3) a third layer of an avidin-biotin complex. Finally, counterstaining was performed, generating biopsy slides with cells positive for peptide YY (PYY), GLP-1, respectively.
  Quantitative real-time polymerase chain reaction (qPCR) : the mRNA expression of the genes of interest glp-1,PYY 3-36 genes as well as the genes used for normalisation 18S were investigated. One biopsy sample from each biopsy site was immediately incubated in RNAlater solution (to preserve mRNA quality) (dna/rna Shield, USA). Subsequently, standard RNA purification, cDNA synthesis and quantitative PCR (qPCR) analysis were performed .
  Interventions: Other: Analyze basal expression incretin for immunolabeling and mRNA expression glucagon-like secretion peptide-1 (GLP-1) and peptide YY (PYY 3-36) incretins by L cells.

INTERVENTIONS:
Other: Analyze basal expression incretin for immunolabeling and mRNA expression glucagon-like secretion peptide-1 (GLP-1) and peptide YY (PYY 3-36) incretins by L cells. — Preoperative and postoperative

SUMMARY:
Prevalence of Obesity and its association with Diabetes Mellitus 2 (DM2) affect a significant percentage of the world's population with great socioeconomic impact, especially for developing countries. Several procedures and interventions are used in its treatment, and the most efficient and with a positive impact on the life of patients with severe obesity and DM2 is Bariatric Surgery.

The objective of is analyze the activity of L cells according to the extension of the bilio-pancreatic loop in T2DM patients undergoing GDYR.

This study 20 adults of both sexes, above 18 years,before and 6 moths after surgery baritric metabolic, randomized the bilio-pancreatic loop in a proportion of 1:1.

Keywords: Roux-en-Y gastroplasty, Immunohistochemistry, L cell, GLP-1, type 2 diabetes.

DETAILED DESCRIPTION:
This is a prospective, randomized (paired) and morphological study involving 20 adult male and female patients (18-65 years) with severe obesity [body mass index (BMI) > 35 kg/m2] and DM2 undergoing Gastroplasty in Diversion Roux-en-Y in the Bariatric and Metabolic Surgery Unit, Department of Gastroenterology, HC-FMUSP, between February 2020 and December 2022. Patients were randomized (https://hcbredcap.com.br/) into two groups of 10 patients each, according to the extension of the bilio-pancreatic loop, in a proportion of 1:1 by computer model. Patients were evaluated preoperatively (T0) and 6 months (T1) after GDYR.

INTRODUTION: Patients with obesity have a suppressed incretin effect and a consequent imbalance of glycemic homeostasis. Bariatric surgery has the potential of T2DM control in up to 90% of patients with severe obesity due to caloric restriction, improvement of insulin resistance, pancreatic beta cell function, and the incretin effect of glycogen-like protein 1.

In this current scenario, metabolic surgery has taken a considerable role in weight loss, contributing to metabolic control, and showing improvement in the state of obesity and related comorbidities. We already know that conservative treatment has been failing 80% of obese patients, while 80% of obese patients who have undergone metabolic surgery are successful in long-term weight loss and resumption of metabolic functionality, showing better results than drug therapy or only lifestyle change 16 . This adaptive procedure, which is aimed at neuroendocrine improvements instead of gastrointestinal restriction and malabsorption 24 , leads to increased serum levels of the incretins (hormones that stimulate a decrease in blood glucose levels) glucagon- like peptide-1 (GLP-1) and peptide YY (PYY 3-36 ) in postprandial patients five years following surgery. They play key roles in stimulating the secretion of insulin by the endocrine pancreas . It is therefore of considerable importance to understand the secretion mechanisms of epithelial intestinal cells as well as the identity and location of cells responsible for the action of these peptides . In the intestinal epithelium we find cells that release incretins to the response of nutrients in contact with intestinal lumen called L cells . L cell found in the distal ileum and large intestine secretes GLP-1 and peptide YY (PYY) promotes they slow gastric emptying and act as a satiety signal to improve glycemic control.

JUSTIFICATION: number of L cells in activity implies better peptide signaling, response and functioning of the neuroendocrine system.

OBJECTIVE: To analize secretion of L cells in the small intestine for immunohistochemistry and mRNA expression levels before and after (6 months) induced by bariatric surgery .

METHODS: Ethic This study was elaborated and will be performed at the Clinical Hospital of the Medical School of the University of São Paulo (HCFMUSP). The patients involved will receive the Informed Consent Form (ICF) for their agreement to participate in the study.

The molecular markers(qRT-PCR) used will be the expression enterohormones themselves by the L cell, that is, GLP-1 and PYY.

The detection of incretin by Immunohistochemical assays, will enable cell labeling and localization, and evidence of cell occurrence/density in portions of the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 to 65 years
* Both sexes
* BMI ≥ 35 kg/m2
* Presence of DM2:
* Glycated Hb ≥ 7.0%
* C-peptide ≥ 3 ng/dl
* Fasting blood glucose ≥ 200 mg/dl (absence of treatment)
* TCLE

Exclusion Criteria:

* Corticosteroid use
* Hepatitis B and C or HIV carriers
* Previous abdominal or bariatric surgery
* Cardiovascular impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-12-05 (Estimated)

PRIMARY OUTCOMES:
Changes number of active L cells | Before and 6 moths after bariatric surgery
  The analysis of the samples of intestinal tract mucosa the patients with DM2 , immunolabeling for GLP-1 and for PYY 3-36 from number of active L cells, before and after bariatric surgery.
Changes mRNA expression levels of active L cells | Before and 6 moths after bariatric surgery
  The analysis of the samples of intestinal tract mucosa from the from patients with DM2 , mRNA expression levels of GLP-1 and PYY 3-36 for active L cells, before and after bariatric surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Aurelio Santo, MD Phd, Principal Investigator — Clinical Hospital of University of Sao Paulo Medical School; Priscila Costa Estabile, MsC, Study Chair — Clinical Hospital of University of Sao Paulo Medical School
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, Brazil

REFERENCES:
- [Background] Miras AD, Kamocka A, Perez-Pevida B, Purkayastha S, Moorthy K, Patel A, Chahal H, Frost G, Bassett P, Castagnetto-Gissey L, Coppin L, Jackson N, Umpleby AM, Bloom SR, Tan T, Ahmed AR, Rubino F. The Effect of Standard Versus Longer Intestinal Bypass on GLP-1 Regulation and Glucose Metabolism in Patients With Type 2 Diabetes Undergoing Roux-en-Y Gastric Bypass: The Long-Limb Study. Diabetes Care. 2021 May;44(5):1082-1090. doi: 10.2337/dc20-0762. Epub 2020 Nov 6. PMID 33158945
- [Background] Estabile PC, Almeida MC, Campagnoli EB, Santo MA, Rodrigues MRDS, Milleo FQ, Artoni RF. IMMUNOHISTOCHEMICAL DETECTION OF L CELLS IN GASTROINTESTINAL TRACT MUCOSA OF PATIENTS AFTER SURGICAL TREATMENT FOR CONTROL OF TYPE 2 DIABETES MELLITUS. Arq Bras Cir Dig. 2022 Jun 17;35:e1651. doi: 10.1590/0102-672020210002e1651. eCollection 2022. PMID 35730880
- [Background] Jorsal T, Rhee NA, Pedersen J, Wahlgren CD, Mortensen B, Jepsen SL, Jelsing J, Dalboge LS, Vilmann P, Hassan H, Hendel JW, Poulsen SS, Holst JJ, Vilsboll T, Knop FK. Enteroendocrine K and L cells in healthy and type 2 diabetic individuals. Diabetologia. 2018 Feb;61(2):284-294. doi: 10.1007/s00125-017-4450-9. Epub 2017 Sep 28. PMID 28956082
- [Background] Guedes TP, Martins S, Costa M, Pereira SS, Morais T, Santos A, Nora M, Monteiro MP. Detailed characterization of incretin cell distribution along the human small intestine. Surg Obes Relat Dis. 2015 Nov-Dec;11(6):1323-31. doi: 10.1016/j.soard.2015.02.011. Epub 2015 Feb 17. PMID 26048514